

# TRIAL STATISTICAL ANALYSIS PLAN

c26502696-01

| BI Trial No.: | 1407-0031 |
|---|---|
| Title: | A phase I, open-label, single-dose trial to investigate metabolism and pharmacokinetics of BI 730357 BS (C-14) administered as oral solution in healthy male volunteers |
| Investigational Product(s): | BI 730357 |
| Responsible trial statistician(s): | |
| | Phone:<br>Fax: |
| | Phone:<br>Fax: |
| Date of statistical analysis plan: | 10 JAN 2019 SIGNED |
| Version: | Final |

**Proprietary confidential information** 

© 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

TSAP for BI Trial No: 1407-0031 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 1. | TA | BLE | $\mathbf{OE}$ | CON | TEN | TC |
|----|----------------|------|---------------|-----|-----|-----|
| 1. | $\mathbf{I} P$ | ADLL | <b>U</b> F | CUN | | 110 |

| TITLE PAGE1 | | |
|---|---|---|
| 1. | TABLE OF CONTENTS. | 2 |
| LIST OF TABLES | | |
| 2. | LIST OF ABBREVIATIONS | 5 |
| 3. | INTRODUCTION | |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | |
| 5. | ENDPOINTS | |
| 5.1 | PRIMARY ENDPOINTS | |
| 5.2 | SECONDARY ENDPOINTS | |
| 5.2.1 | Key secondary endpoints | |
| 5.2.2 | Secondary endpoints | |
| 6. | GENERAL ANALYSIS DEFINITIONS | 11 |
| 6.1 | TREATMENT | |
| 6.2 | IMPORTANT PROTOCOL DEVIATIONS | |
| 6.3 | SUBJECT SETS ANALYSED. | |
| 6.5 | POOLING OF CENTRES | 13 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS | |
| 7. | PLANNED ANALYSIS | 15 |
| 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION | 16 |
| 7.3 | TREATMENT COMPLIANCE | 16 |
| <b>7.4</b> | PRIMARY ENDPOINTS | |
| 7.5 | SECONDARY ENDPOINTS | |
| 7.5.1 | Key secondary endpoint | |
| 7.5.2 | Secondary endpoints | 17 |
| 7.7 | EXTENT OF EXPOSURE | 17 |
| 7.8 | SAFETY ANALYSIS | |
| 7.8.1 | Adverse events | |
| 7.8.2 | Laboratory data | |
| 7.8.3 | Vital signs | |

# Boehringer Ingelheim TSAP for BI Trial No: 1407-0031

**10.** 

| <b>TSAP</b> | for BI Trial No: 1407-0031 ry confidential information © 2019 Boehringer Ingelheim Internation | |
|---|---|---|
| Proprietar | ry confidential information © 2019 Boehringer Ingelheim Internation | al GmbH or one or more of its affiliated companies |
| 7.8.4 | ECG | 20 |
| 7.8.5 | Others | 20 |
| 8. | REFERENCES | 21 |

HISTORY TABLE......23

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1407-0031 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# LIST OF TABLES

| Table 6.1: 1 | Flow chart of analysis phases for statistical analyses of AEs, safety | |
|---|---|---|
| | laboratory data and vital signs | 11 |
| Table 6.2: 1 | Important protocol deviations | 12 |
| Table 6.3: 1 | Subject sets analysed | 13 |
| Table 10: 1 | History table | 23 |

TSAP for BI Trial No: 1407-0031 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### LIST OF ABBREVIATIONS 2.

| Term | Definition / description |
|---|---|
| ADPC | Proper name of the analysis dataset containing PK concentrations per time-point or per time-interval |
| ADPP | Proper name of the analysis dataset containing calculated PK parameters |
| ADS | Analysis dataset |
| AE | Adverse Event |
| AESI | Adverse event of special interest |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| $AUC_{0\text{-tz}}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point |
| BI | Boehringer Ingelheim |
| BLQ | Below the lower limit of quantification |
| BMI | Body Mass Index |
| BP | Blood Pressure |
| BRPM | Blinded Report Planning Meeting |
| $C_{max}$ | Maximum measured concentration of the analyte in plasma |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| CV | Arithmetic coefficient of variation |
| ECG | Electrocardiogram |
| EDC | Electronic Data Capture |
| FAS | Full Analysis Set |
| fe <sub>faeces</sub> , 0-t2 | fraction of [14C]-radioactivity excreted in faeces as percentage of the administered dose over the time interval from 0 to to $t_2$ (where $t_{2 is}$ the last quantifiable data point across all subjects) |
| fe <sub>urine, 0-t2</sub> | fraction of [14C]-radioactivity excreted in urine as percentage of the administered dose over the time interval from 0 to $t_2$ (where $t_{2 is}$ the last quantifiable data point across all subjects) |
| gCV | geometric coefficient of variation |
| gMean | Geometric mean |
| ICH | International Conference On Harmonisation |
| IPD | Important Protocol Deviation |

TSAP for BI Trial No: 1407-0031 
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|--------|----------------------------------------------|
| LLOQ | Lower limit of quantification |
| MedDRA | Medical Dictionary For Regulatory Activities |
| NOA | Not analysed |
| NOP | No peak detectible |
| NOR | No valid result |
| NOS | No sample available |
| PK | Pharmacokinetics |
| PKS | Pharmacokinetic parameter set |
| PR | Pulse Rate |
| PT | Preferred Term |
| Q1 | Lower Quartile |
| Q3 | Upper Quartile |
| SA | Statistical Analysis |
| SD | Standard Deviation |
| SOC | System Organ Class |
| TCM | Trial Clinical Monitor |
| ToC | Table of Contents |
| TMW | Trial Medical Writer |
| TS | Treated Set |
| TSAP | Trial Statistical Analysis Plan |
| ULN | Upper limit of normal range |

TSAP for BI Trial No: 1407-0031

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 3. INTRODUCTION

As per ICH E9 (1), the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This TSAP assumes familiarity with the CTP, including Protocol Amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomization.

Study data will be stored in a trial database within the Medidata Rave system.

The statistical analyses will be performed within the validated working environment CARE, including SAS<sup>TM</sup> (current Version 9.4, by SAS Institute Inc., Cary, NC, USA), and a number of SAS<sup>TM</sup>-based tools (e.g., macros for the analyses of AE data or laboratory data; Report Appendix Generator system (RAGe) for compilation/formatting of the CTR appendices).

PK parameters will be calculated using Phoenix WinNonlin<sup>TM</sup> software (version 6.3, Certara USA Inc., Princeton, NJ, USA).

#### CHANGES IN THE PLANNED ANALYSIS OF THE STUDY 4.

All analyses described in this TSAP are in accordance with the statistical methods described in the CTP.

TSAP for BI Trial No: 1407-0031

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 5. ENDPOINTS

### 5.1 PRIMARY ENDPOINTS

Primary endpoints are PK endpoints of mass balance recovery of [14C]-radioactivity as defined in Section 5.5.1.1 of the CTP:

- fe<sub>urine, 0-t2</sub> (fraction of [<sup>14</sup>C]-radioactivity excreted in urine as percentage of the administered dose over the time interval from 0 to t<sub>2</sub> (where t<sub>2</sub> is the last quantifiable data point across all subjects))
- fe<sub>facces, 0-t2</sub> (fraction of [<sup>14</sup>C]-radioactivity excreted in facces as percentage of the administered dose over the time interval from 0 to t<sub>2</sub> (where t<sub>2</sub> is the last quantifiable data point across all subjects))

**CTP**: Timeframe: The timeframe for determination of these endpoints depends on excretion/recovery of radioactivity and may vary between 2-7 weeks, inclusive, after drug administration.

#### 5.2 SECONDARY ENDPOINTS

#### 5.2.1 Key secondary endpoints

Not applicable

## 5.2.2 Secondary endpoints

Secondary PK endpoints will be defined as in Section 5.5.1.2 of the CTP for [<sup>14</sup>C]-radioactivity and BI 730357 in plasma:

- C<sub>max</sub> (maximum measured concentration of the analyte)
- AUC<sub>0-tz</sub> (area under the concentration-time curve of the analyte over the time interval from 0 to the last quantifiable time point)

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1407-0031 
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1407-0031

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENT

For basic study information on treatments to be administered, assignments of dose groups, and selection of doses, cf. Section 4 of the CTP.

All subjects were planned to be treated with a single dose of 50 mg BI 730357 BS (C-14) (BI 730357 mixed with [C-14]BI 730357 BS)

For statistical analysis of AEs, safety laboratory data and vital signs, the following analysis phases are defined for each subject:

Table 6.1: 1 Flow chart of analysis phases for statistical analyses of AEs, safety laboratory data and vital signs

| Study analysis phase | Label | Start (inclusive) | End (exclusive) |
|---|---|---|---|
| Screening | Screening | Date of informed consent | Date/time of administration of study drug |
| On-treatment | BI 730357 | Date/time of administration of study drug | 12:00 a.m. on day after end<br>of REP<br>(REP ends 7 days after date<br>of administration of study<br>drug) |
| Follow-up | F/U | 12:00 a.m. on day after end of REP | 12:00 a.m. on day after trial completion date |

CTR Section 15, Appendix 16.1.13.1.8.2 and Appendix 16.1.13.1.8.3 AE displays will present results for the on-treatment phase only. Appendix 16.1.13.1.8.1 will present results for the screening, on-treatment and follow-up phase.

Additionally, the following total will be provided in CTR Section 16.1.13.1.8.1 AE tables:

• "Total", defined as the total over all study phases (incl. screening, on-treatment, and follow-up)

#### 6.2 IMPORTANT PROTOCOL DEVIATIONS

Consistency check listings (for identification of violations of time windows) and a list of protocol deviations (e.g. deviations in drug administration, in blood sampling times, etc.) will be provided to be discussed at the RPM/DBLM. At this meeting, it will be decided whether a discrepant data value can be used in analyses or whether it must be corrected in the clinical database. Each protocol deviation must be assessed to determine whether it is an IPD. For definition of IPDs, and for the process of identification of these, refer to the BI reference document "Identify and Manage Important Protocol Deviations (iPD)" (2).

If any IPDs are identified, they are to be summarised into categories and will be captured in the RPM/DBLM minutes via an Excel spreadsheet (3). The table below contains the categories which are considered to be IPDs in this trial. If the data show other IPDs, this table will be supplemented accordingly by the time of the RPM/DBLM.

IPDs will be summarised and listed.

TSAP for BI Trial No: 1407-0031

Table 6.2: 1 Important protocol deviations

| Cat<br>/ Co | egory | Description |
|---|---|---|
| A | | Entrance criteria not met |
| | A1 | Inclusion criteria violated |
| | A2 | Exclusion criteria violated |
| В | | Informed consent |
| | B1 | Informed consent not available |
| | B2 | Informed consent too late |
| C | | Trial medication and randomisation |
| | C1 | Non-compliance |
| | C2 | Incorrect dose of trial medication |
| D | | Concomitant medication |
| | D1 | Prohibited medication use |
| E | | Missing data |
| | | None <sup>1</sup> |
| G | | Other trial specific important violations |
| | G1 | Certain violations of procedures used to measure primary or secondary PK data |

Deviations C1, C2 and G1 can only be detected at the trial site.

Source: BI reference document "Identify and Manage Important Protocol Deviations (iPD)" (2).

#### 6.3 SUBJECT SETS ANALYSED

All entered subjects who received study medication will be included in the safety analysis and in the PK analysis depending on the availability of measurement values, and on their adherence to the CTP.

The following subject sets will be defined for statistical analysis:

- Treated set (TS):
  - This subject set includes all subjects who were documented to have received one dose of study drug. This is the full analysis set population in the sense of ICH-E9. It will be used for analysis of safety, demographic data and baseline characteristics.
- Pharmacokinetic parameter analysis set (PKS):
  This subject set includes all subjects in the TS who provide at least one value for primary or secondary PK parameter that was not excluded because of iPDs relevant to

<sup>&</sup>lt;sup>1</sup> Missing visits, evaluations, and tests will be considered missing data, not IPDs

TSAP for BI Trial No: 1407-0031

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

the statistical evaluation of PK endpoints as defined in Section 7.3 of the CTP. The discussion of all exceptional cases and problems and the decisions on the allocation of subjects to analysis sets will be made at latest at the RPM/DBLM

Table 6.3: 1 Subject sets analysed

| | Subject set | |
|---------------------------|-------------|-----|
| Class of endpoint | TS | PKS |
| Disposition | X | |
| Exposure | X | |
| IPDs | X | |
| Demographic/baseline data | X | |
| Safety parameters | X | |
| Primary PK endpoints | | X |
| Secondary PK endpoints | | X |
| Further PK endpoints | | X |

### 6.5 POOLING OF CENTRES

This section is not applicable, because the study was performed in only one centre.

#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Data of screened subjects who were withdrawn from the trial prior to first administration of any study drug will not be reported in the CTR.

Data of subjects who failed to complete all periods of the study (dropouts or withdrawals) will be reported in the CTR as far as their data are available. All withdrawals will be documented and the reason for withdrawal recorded in the CTR.

**CTP**: With respect to safety evaluations, it is not planned to impute missing values.

The only exception where imputation might be necessary for safety evaluation are AE dates. Missing or incomplete AE dates are imputed according to BI standards (4) [001-MCG-156 RD-01].

Missing data and outliers of PK data are handled according to BI standards (5).

Blood/ Plasma/ Urine/ Faeces drug concentration or [14C]-radioactivity-time profiles

**CTP**: Drug concentration data identified with NOS (no sample available), NOR (no valid result), NOA (not analysed), BLQ (below the lower limit of quantification), or NOP (no peak detectable) will be displayed as such and not replaced by zero at any time point (this rule also applies also to the lag phase, including the predose values).

#### Pharmacokinetic parameters

**CTP**: For the non-compartmental analysis, concentration data identified with NOS, NOR or NOA will generally not be considered. Concentration values in the lag phase identified as BLQ or NOP will be set to zero. All other BLQ/NOP values of the profile will be ignored. The lag phase is defined as the period between time zero and the first time point with a concentration above the quantification limit.

## 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

The last non-missing value determined prior to the first study drug administration will be defined as baseline.

Time windows are defined in Section 6.1 of the CTP. Adherence to time windows will be checked at the RPM/DBLM.

#### 7. PLANNED ANALYSIS

The format of the listings and tables will follow the BI guideline "Reporting of clinical trials and project summaries" ( $\underline{6}$ ).

The individual values of all subjects will be listed, sorted by dose group, subject number and visit. AE listings will be sorted by assigned treatment (see Section 7.8.1 below for details). The listings will be contained in Appendix 16.2 (SDL) of the CTR.

The following standard descriptive statistical parameters will be displayed in summary tables of continuous variables:

N number of non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Median median Max maximum

For plasma concentrations as well as for all PK parameters, the following descriptive statistics will additionally be calculated:

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

The data format for descriptive statistics of plasma concentrations will be identical with the data format of the respective concentrations. The descriptive statistics of PK parameters will be calculated using the individual values with the number of decimal places as provided by the evaluation program. Then the individual values as well as the descriptive statistics will be reported with three significant digits in the CTR.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment. Percentages will be rounded to one decimal place. The category missing will be displayed if and only if there actually are missing values. Percentages will be based on all subjects in the respective subject set whether they have non-missing values or not.

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the report. These will be based on the TS.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Concomitant diseases will be coded according to MedDRA, version 21.1. Concomitant medication will be coded according to the World Health Organisation – Drug Dictionary, version of March 2018.

Only descriptive statistics are planned for this section of the report.

A medication will be considered concomitant to a dose group, if it

- is ongoing at the time of first administration of this treatment, or
- starts within the analysis phase of the respective treatment (see <u>Section 6.1</u> for a definition of treatments and analysis phases).

#### 7.3 TREATMENT COMPLIANCE

Treatment compliance will not be analysed as a specific endpoint (cf. Section 5.4.2). Any deviations from complete intake will be addressed in the RPM/DBLM (cf. Section 6.2) and described in the CTR.

#### 7.4 PRIMARY ENDPOINTS

Only descriptive statistics are planned for this section of the CTR. These will be based on the PKS. The analysis of standard PK parameters is performed according to BI standards (5) [001-MCS-36-472 RD-01].

### Exclusion of PK parameters

The ADS ADPP contains column variables APEXC and APEXCO indicating inclusion/exclusion (APEXC) of a PK parameter and an analysis flag comment (APEXCO). All analyses based on the PKS are based on PK parameter values which are not flagged for exclusion, i.e. with APEXC equal to "Included".

#### Exclusion of plasma/urine concentrations

The ADS ADPC (PK concentrations per time-point or per time-interval) contains column variables ACEXC or ACEXCO indicating inclusion/exclusion (ACEXC) of a concentration and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to "ALL CALC", the value will be excluded for all types of analyses based on concentrations. If ACEXCO is set to "DESC STATS" the value will be excluded from descriptive evaluations per planned time point/time interval. If ACEXCO contains the addition "TIME VIOLATION" or "TIME DEVIATION", the value can be used for further analyses based on actual times. If ACEXCO is set to "HALF LIFE", the value will be excluded from half-life calculation only; the value is included for all other analyses. Excluded concentration itself will be listed in the CTR associated with an appropriate flag.

Further details are given in "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies" (5) and "Description of Analytical Transfer Files and PK/PD Data Files" (7).

#### 7.5 SECONDARY ENDPOINTS

#### 7.5.1 Key secondary endpoint

This section is not applicable as no key secondary endpoint has been specified in the CTP.

#### 7.5.2 Secondary endpoints

Secondary PK endpoints will be assessed descriptively. This will be based on the PKS. The analysis of standard PK parameters is performed according to BI standards (5) [001-MCS-36-472 RD-01].

See <u>Section 7.4</u> of this TSAP for details regarding exclusion of PK parameters and plasma concentrations.

## 7.7 EXTENT OF EXPOSURE

Treatment exposure will only be listed by means of the date and time of drug administration.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the TS.

#### 7.8.1 Adverse events

AEs will be coded with the most recent version of MedDRA.

The analyses of AEs will be descriptive in nature. All analyses of AEs will be based on the number of subjects with AEs and not on the number of AEs.

For analysis, multiple AE occurrence data on the electronic case report form (eCRF) will be collapsed into an AE event provided that all of the following applies:

- All AE attributes are identical (LLT, intensity, action taken, therapy required, seriousness, reason for seriousness, relationship, outcome, AESI)
- The occurrences were time-overlapping or time-adjacent (time-adjacency of two occurrences is given if the second occurrence started at most 1 hour after the first occurrence ended).

For further details on summarization of AE data, please refer to "Analysis and presentation of adverse event data from Clinical Trials" (8) and "Handling of missing and incomplete AE dates" (4).

The analysis of AEs will be based on the concept of treatment emergent AEs. That means that all AEs will be assigned to the screening or treatment phases as defined in <u>Section 6.1</u>. AEs will be analysed based on actual treatments, as defined in <u>Table 6.1: 1</u>.

An overall summary of AEs will be presented. This overall summary will comprise summary statistics for the class of other significant AEs according to ICH E3 and for the class of AESIs.

**CTP:** *The following are considered as AESIs:* 

- Hepatic injury

  A hepatic injury is defined by the following alterations of hepatic laboratory
  parameters:
  - o an elevation of AST (aspartate transaminase) and/or ALT(alanine transaminase)  $\geq$ 3-fold ULN combined with an elevation of total bilirubin  $\geq$ 2-fold ULN measured in the same blood sample, or
  - o aminotransferase (ALT, and/or AST) elevations  $\geq$ 10 fold ULN
- Severe infections (according to RCTC grading)
- Opportunistic and mycobacterium tuberculosis infections

The investigator had to classify on the eCRF whether an observed AE was an AESI or not.

According to ICH E3 (9), AEs classified as 'other significant' need to be reported and will include those non-serious and non-significant AEs

- (i) which are marked haematological or other lab abnormalities, or
- (ii) which were reported with 'action taken with study treatment' other than 'dose not changed', or
- (iii) which lead to significant concomitant therapy as identified by the Clinical Monitor/Investigator at a Medical Quality Review Meeting.

The frequency of subjects with AEs will be summarised by treatment, primary system organ class and preferred term. AEs which were considered by the investigator to be drug related will be summarised separately. Separate tables will also be provided for subjects with SAEs, subjects with AESIs and subjects with other significant AEs (according to ICH E3 (9)). AEs will also be summarized by maximum intensity.

The system organ classes will be sorted by total frequency, preferred terms will be sorted by total frequency (within system organ class).

For disclosure of AE data on ClinicalTrials.gov, the frequency of subjects with non-serious AEs occurring with an incidence of greater than 5 % (in preferred terms) will be summarised by treatment, primary SOC and preferred term. The frequency of subjects with SAEs will also be summarised.

For disclosure of AE data in the EudraCT register, the frequency of AEs, the frequency of non-serious AEs with an incidence of greater than 5 % (in preferred terms) and the frequency of SAEs will be summarised.

For support of lay summaries, the frequency of subjects with drug-related SAEs will be summarised by treatment, primary system organ class and preferred term.

#### 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standard "Display and Analysis of Laboratory Data" (10). Alpha-1 Acid Glycoprotein values will only be listed.

Analyses will be based on normalised values, which means transforming to a standard unit and a standard reference range.

Descriptive statistics of laboratory values over time and for the difference from baseline (see <u>Section 6.7</u>) will be provided. Frequency tables of changes between baseline and last value on treatment with respect to the reference range will be presented.

Unscheduled measurements of laboratory data will be assumed to be repeat measurements of the most recent scheduled measurement (e.g. for follow-up or confirmation of a particular value). Therefore, unscheduled measurements will be assigned to the planned time point of the previous scheduled measurement. Descriptive statistics will be calculated by planned time point based on the worst value of the subject at that planned time point (or assigned to that planned time point).

Possibly clinically significant abnormal laboratory values are only those identified either in the Investigator's comments on the eCRF or at the RPM/DBLM at the latest. It is the Investigator's responsibility to decide whether a lab value is clinically significant abnormal or not. Standard or project-specific rules for flagging clinically significant values will not be applied in this study.

Clinically relevant findings in laboratory data will be reported as AEs and will be analysed as part of AE analysis.

## 7.8.3 Vital signs

The analysis of vital signs will be descriptive in nature. Descriptive statistics of vital signs over time and for the difference from baseline (see Section 6.7) will be provided.

Unscheduled measurements of vital signs will be assigned to planned time points in the same way as described above for laboratory data. However, for vital signs, descriptive statistics will be calculated by planned time point based on the last value of the subject at that planned time point (or assigned to that planned time point).

Clinically relevant findings in vital signs data will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analysed as such.

#### 7.8.4 ECG

Abnormal findings in 12-lead ECG will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analysed as such. No separate listing or analysis of ECG data will be prepared.

### **7.8.5** Others

Physical examination findings will be reported as relevant medical history/baseline condition (i.e., a condition already existent before intake of first study drug) or as AE and will be summarised as such. No separate listing or analysis of physical examination findings will be prepared.

TSAP for BI Trial No: 1407-0031 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 8. **REFERENCES**

| 1. | CPMP/ICH/363/96: "Statistical Principles for Clinical Trials", ICH Guideline Topic E9, Note For Guidance on Statistical Principles for Clinical Trials, current version |
|---|---|
| 2. | 001-MCS-40-413_1.0: "Identify and Manage Important Protocol Deviations (iPD)", current version; IDEA for CON |
| 3. | "Template Domain DV", current version; Section "Resources and Key User Emails" on ICBI homepage |
| 4. | 001-MCG-156_RD-01: "Handling of missing and incomplete AE dates", current version; IDEA for CON |
| 5. | 001-MCS-36-472_RD-01: "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies", current version; IDEA for CON |
| 6. | 001-MCG-159: "Reporting of Clinical Trials and Project Summaries", current version; IDEA for CON |
| 7. | 001-MCS-36-472_RD-03: "Description of Analytical Transfer Files and PK/PD Data Files", current version; IDEA for CON |
| 8. | 001-MCG-156: "Analysis and Presentation of Adverse Event Data from Clinical Trials", current version; IDEA for CON |
| 9. | CPMP/ICH/137/95: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version |
| 10. | 001-MCG-157: "Display and Analysis of Laboratory Data", current version; IDEA for CON |

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1407-0031 
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **10. HISTORY TABLE**

Table 10: 1 History table

| Version | Date | Author | Sections | Brief description of change |
|---|---|---|---|---|
| | (DD-MMM-YY) | | changed | |
| Final | 10-JAN-2019 | | None | This is the final TSAP without any |
| | | _ | | modification |